CLINICAL TRIAL: NCT03545568
Title: Sialic Acid Supplementation in NANS Deficiency: An Open-label, Proof of Concept, Two-centers Study
Brief Title: Sialic Acid Supplementation in N-Acetylneuraminic Acid Synthase (NANS) Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Christel Tran, Principal investigator, University of Lausanne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-00284
Record Dates: First submitted 2018-05-08; First posted 2018-06-04 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-05

CONDITIONS: N-Acetylneuraminic Acid Storage Disease
Keywords: Sialic acid; Monosaccharide
MeSH Terms: conditions — N-Acetylneuraminic acid storage disease

STUDY DESIGN:
Intervention Model Description: Open label individual patient clinical trial study of small sample size
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: sialic acid (Other)
  Interventions: Other: Neu5Ac supplementation

INTERVENTIONS:
Other: Neu5Ac supplementation — Sialic acid as N-Acetyl-neuraminic acid dehydrate (Neu5Ac) 150 mg/kg/d (max 12g/d) in three doses orally in subjects with NANS deficiency compared to controls

SUMMARY:
This study is aimed at assessing the impact of short-term (3 days) exogenous sialic acid supplementation on endogenous biomarkers of sialic acid metabolism in NANS deficient patients.

DETAILED DESCRIPTION:
NANS deficiency is a genetic disorder presenting clinically with intellectual development disorder, skeletal dysplasia and dysmorphic features. It has recently been described in 9 patients (4 children and 5 adults). Biallelic mutations in the NANS (N-Acetylneuraminic acid synthase) gene cause a block in the endogenous synthesis of sialic acid and accumulation of the precursor, N-acetyl mannosamine (ManNAc). In a cell culture model, this block results in hyposialylation of glycoproteins and glycolipids. It seems likely that in human, this enzyme deficiency impairs the sialylation of glycolipids and glycoproteins, known to be essential for brain development. Exogenously added sialic acid partially rescued the phenotype of NANS-deficient zebra fish. Currently there is no approved treatment for patients with NANS deficiency. The investigators concluded that exogenous sialic acid supplementation might be useful for NANS patients. Given that sialic acid is found as both, a free sugar and in a bound form in standard nutrition as well as in high quantities in breast milk, it can be considered as a safe nutritional ingredient; this notion is fully supported by animal toxicity studies.

The use of sialic acid in NANS deficiency is in line with oral supplementation of specific sugars for treatment of other glycosylation and sialylation defects such as congenital disorders of glycosylation (CDG) and myopathy with mutation in the gene GNE. This novel monosaccharide therapy represents an opportunity to address fundamental biochemical questions about the relative contribution of endogenous and dietary sources on sialic acid metabolism and its potential role as a future therapy for NANS patients.

ELIGIBILITY:
Inclusion Criteria for controls:

* 4 healthy adults aged 18 to 60 years (inclusion in Switzerland)

Inclusion Criteria for subjects with NANS deficiency:

* 4 adults aged 18 to 60 years with genetically proven NANS deficiency (inclusion in Italy)
* 2 children aged 1 to 18 years with genetically proven NANS deficiency (inclusion in Switzerland)

Exclusion Criteria for controls:

* Medication, Restrictive diet (e.g. lactose free diet), obesity or other co-morbidities (e.g. neurological disease, developmental delay)

No exclusion Criteria for subjects

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Metabolite concentration | -30 min before ingestion of Neu5Ac at day 2. 120 min, 240 min and 360 min after Neu5Ac ingestion at day 2. 120 min after neu5Ac ingestion at day 3-4. With no Neu5Ac supplementation at day 5
  The primary endpoint is the change of metabolite concentration after N-Acetyl-D neuraminic acid (Neu5Ac) supplementation from day 2 to day 4 and follow-up visit at day 5

SECONDARY OUTCOMES:
Urine and plasma concentrations of N-acetyl mannosamine (ManNAc) | 30 min before ingestion of Neu5Ac at day 2. 120 min, 240 min and 360 min after Neu5Ac ingestion at day 2. 120 min after neu5Ac ingestion at day 3-4. With no Neu5Ac supplementation at day 5
  Change in ManNAc concentration from baseline and after exogenous sialic acid supplementation
Urine and plasma concentrations of free sialic acid | 30 min before ingestion of Neu5Ac at day 2. 120 min, 240 min and 360 min after Neu5Ac ingestion at day 2. 120 min after neu5Ac ingestion at day 3-4. With no Neu5Ac supplementation at day 5
  Change in free sialic acid concentration from baseline and after exogenous sialic acid supplementation
Urine and plasma concentrations of total sialic acid | 30 min before ingestion of Neu5Ac at day 2. 120 min, 240 min and 360 min after Neu5Ac ingestion at day 2. 120 min after neu5Ac ingestion at day 3-4. With no Neu5Ac supplementation at day 5
  Change in total sialic acid concentration from baseline and after exogenous sialic acid supplementation
Urine and plasma concentrations of N-Acetyl-D neuraminic acid (Neu5Ac) | 30 min before ingestion of Neu5Ac at day 2. 120 min, 240 min and 360 min after Neu5Ac ingestion at day 2. 120 min after neu5Ac ingestion at day 3-4. With no Neu5Ac supplementation at day 5
  Change in Neu5Ac concentration from baseline and after exogenous sialic acid supplementation
Urine and plasma metabolomic profile | 30 min before ingestion of Neu5Ac at day 2. 120 min, 240 min and 360 min after Neu5Ac ingestion at day 2. 120 min after neu5Ac ingestion at day 3-4. With no Neu5Ac supplementation at day 5
  Change in metabolomic profile from baseline and after exogenous sialic acid supplementation
Blood pressure in mmHg | -30 min before Neu5Ac ingestion at day 2 to 4. With no Neu5Ac supplementation at day 5
  Measure of blood pressure (mmHg) supplementation
Heart beat per minute (BPM) | -30 min before Neu5Ac ingestion at day 2 to 4. With no Neu5Ac supplementation at day 5
  Measure of heart BPM at baseline and after exogenous sialic acid supplementation
Body weight (kg) | -30 min before Neu5Ac ingestion at day 2 to 4. With no Neu5Ac supplementation at day 5
  Measure of body weight at baseline and after exogenous sialic acid supplementation
Dietary parameters | 1x/day from day 1 to day 5 (end of the study)
  A self-reporting daily dietetic diary will be recorded for each participant.

CONTACTS AND LOCATIONS:
Locations (2):
- Struttura Semplice Dipartimentale di Genetica Clinica, Reggio Emilia, Italy
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No